CLINICAL TRIAL: NCT06134453
Title: The Effect of Reiki on Surgical Fear and Anxiety
Brief Title: Evaluation of the Effect of Reiki on Surgical Fear and Anxiety in Laparoscopic Cholecystectomy; Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hamide Sisman, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS312
Record Dates: First submitted 2023-08-06; First posted 2023-11-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Supportive Care
Keywords: Cholecystectomy; Surgical Fear; Surgical Anxiety; Reiki
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Reiki, Sham Reiki, Control Group
Who Masked: Participant
Masking Description: Sham reiki will be applied by a nurse who has not received reiki training. He will hold his hands in accordance with the Reiki protocol in the specified chakra areas of the patient for the specified time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki (Experimental): According to randomization, patients in the reiki group will be taken to a quiet single room and reiki will be applied for approximately 25-30 minutes. Reiki practice will be applied by a researcher who has been trained at the Reiki Master level.
  Interventions: Other: Reiki/Sham Reiki
- Sham Reiki (Sham Comparator): According to randomization, the patients in the sham reiki group were taken to a quiet single room and sham reiki was applied for approximately 25-30 minutes. will be applied. According to random distribution, patients in the sham reiki group will be taken to a quiet single room and sham reiki will be applied for approximately 25-30 minutes. Sham Reiki will be administered by a healthcare professional who has not received Reiki training. Their hands will remain in the same position and for the same duration as if they were actually doing Reiki, but Reiki energy will not be given to the patient.
  Interventions: Other: Reiki/Sham Reiki
- Control Group (No Intervention): The control group will be given routine care in the pre-operative waiting room without any intervention, and the data collection tools will be applied at the same time as the experimental group, twice at 30-minute intervals.

INTERVENTIONS:
Other: Reiki/Sham Reiki — Reiki will be applied to the patients by the research nurse who is at the Reiki master level. Sham Reiki will remain in the same position and for the same duration as if Reiki was performed by a healthcare professional who has not received Reiki training, but Reiki energy will not be given to the patient. No intervention will be made to the control group.
  Other Names: Control Group
  Arms: Reiki; Sham Reiki

SUMMARY:
surgical intervention; It is defined as an emergency or planned treatment method for the purpose of diagnosis, treatment and symptom reduction in cases of deformity, injury, and disease with hands and tools. Although these interventions are practices aimed at protecting life, whether it is large or small, urgent or planned, it is both physiological and psychological trauma for the patient. The decision of surgical intervention may cause anxiety in individuals regardless of the type of surgical procedure. Fear of anesthesia, fear of death, possibility of postoperative complications, pain, changes in activities of daily living, loss of social life and loss of control may cause anxiety. Reiki, a complementary and alternative medicine (CAM) method, is a bioenergy based on the body's energy use and has been used for centuries in the prevention and treatment of certain diseases in various cultures. Reiki is thought to help balance the body's natural energy systems and reduce anxiety by transferring existing energy through the hands. Studies on the effectiveness of reiki, which is increasingly used worldwide and recommended as a treatment approach in health care, are insufficient. The aim of this study, which was planned as a three-group interventional randomized control, was to evaluate the effect of reiki on surgical fear and anxiety of patients who will undergo laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The results of the power analysis using the Gpower 3.1.9.2 program, it was planned to have 16 patients in reiki, 16 patients in sham reiki, and 16 patients in the control group, and study groups were determined by simple randomization method. The research data were collected between November 2022 and September 2023 in the operating room waiting room, in a quiet single room. Pre-application, "Personal Information Form", "Surgical Fear Form" and Surgical Anxiety Form" was applied to 12 patients who met the study criteria with the permission of the ethics committee. Data were collected in the operating room waiting room before and after Reiki. After obtaining the patient's consent, the Personal Information Form, the Surgical Fear Scale, and the Surgical Anxiety Scale were applied and recorded. According to randomization, the patients in the reiki/sham reiki group were taken to a quiet single room, and reiki/sham reiki was applied for approximately 25-30 minutes. Reiki application was applied by a researcher who received Reiki Master level training, and sham Reiki was applied by a health professional who did not receive Reiki training. A written protocol is provided to both the Reiki practitioner and Sham Reiki practitioner describing hand positions, areas of practice, sequence, and times. The "Surgical Fear Scale" and "Surgical Anxiety Scale" were applied again 5 minutes after the end of the application. In the control group according to randomization. The "Personal Information Form" was recorded by applying the "Surgical Fear Scale" and the "Surgical Anxiety Scale". 30 minutes of the evaluation were recorded by repeating the "Surgical Fear Scale" and "Surgical Anxiety Scale".

ELIGIBILITY:
Inclusion Criteria:

* 18-65 age range,
* No vision-hearing problem,
* Able to communicate verbally
* No diagnosed psychiatric problem,
* No history or current history of substance use,
* will receive general anesthesia,
* ASA I, II
* Laparoscopic cholecystectomy was planned,

Exclusion Criteria:

* Patients who develop a serious complication after surgery (patients who may need respiratory support and close monitoring due to metabolic disorders, hypothermia, or hemodynamic instability)
* Patients who have previously received energy therapies such as Reiki Touch Therapy / Therapeutic Touch / Healing Touch

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Comparison of participants' surgical fear mean scores before and after Reiki application | [Time Frame: day 0]
  In the "Surgical Fear Scale", the lowest score that can be obtained from the subscales is 0 and the highest score is 40. The lowest score of the scale is 0 and the highest is 80. A high score indicates that fear is high.
Comparison of participants' "Surgical Anxiety Scale" average scores before and after Reiki application | [Time Frame: day 0]
  "The highest score that can be obtained from the Surgical Anxiety Scale is 80, and the lowest score is 20. The higher the total anxiety score, the higher the person's anxiety level is interpreted.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A decision will be made after the study is completed.